CLINICAL TRIAL: NCT02251782
Title: Adherence to Minimally Invasive CRC Screening In Non-Adherent Patients Who Have Not Completed Colorectal Cancer Screening
Brief Title: Adherence to Minimally Invasive Testing
Acronym: ADMIT
Status: Completed | Type: Observational
Sponsor: Epigenomics, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: SPR 0026
Record Dates: First submitted 2014-09-24; First posted 2014-09-29 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Epi proColon Group: Subjects assigned to the Epi proColon Group will be offered the Epi proColon test for colorectal cancer screening.
  Interventions: Device: Epi proColon Test
- FIT Group: Subjects in the FIT Group will be offered a fecal immunochemical test (FIT test) for colorectal cancer screening.
  Interventions: Device: Fecal Immunochemical Test (FIT)
- Usual Care Group: For the purpose of comparison to usual care, participating health systems will build an anonymized group of patients meeting study eligibility criteria, who do not participate in the study. This group will serve as a passive control and their CRC screening activity will be monitored via Medical Record.

INTERVENTIONS:
Device: Epi proColon Test — Subjects assigned to the Epi proColon arm will receive information on the Epi proColon test outlined in a template script. They will then be offered a blood draw for Epi proColon testing. The blood draw can be fulfilled at the clinic or at a specified blood draw station, at the convenience of the patient. Epi proColon plasma samples will be sent to a central laboratory for testing. If no test result is recorded within 4 weeks, patients will be mailed a reminder to complete testing. If no result is recorded within 2 weeks of the mailed reminder, subjects will be recorded as non-adherent to screening. Subjects with negative test results will be mailed a notice of result and reminder to continue screening. Subjects with positive tests will be contacted and counseled to undergo colonoscopy.
  Groups: Epi proColon Group
Device: Fecal Immunochemical Test (FIT) — Subjects assigned to the FIT arm will receive information on the FIT test outlined in a template script. They will then be provided a FIT kit to take home and asked to send a stool sample to the testing lab following the kit instructions. If no test result is recorded within 4 weeks, subjects will receive a mailed reminder to complete testing. If no result is recorded within 2 weeks of the mailed reminder, subjects will be recorded as non-adherent to screening. Subjects with negative test results will be mailed a notice of result and reminder to continue screening. Subjects with positive tests will be contacted and counseled to undergo colonoscopy.
  Groups: FIT Group

SUMMARY:
Colorectal cancer (CRC) screening has been demonstrated to reduce long term disease burden and costs. Unfortunately, less than 65 % of age-eligible persons in the US are actually screened for CRC. The leading methods, colonoscopy and FIT (fecal immunochemical test) testing, both have patient-associated barriers that reduce their use. The combination of bowel preparation and procedure time are barriers to colonoscopy, while stool handling as part of the sampling protocol reduces FIT usage.

It has been hypothesized and supported by a variety of preference studies that the availability of a blood-based assay for CRC screening would increase patient participation and adherence to CRC screening by reducing barriers that prevent participation.

This study is designed to investigate the relative participation in CRC screening in average risk, screening eligible patients with demonstrated non-adherence to guideline-recommended screening modalities. Participation with the fecal immunochemical test (FIT) and the blood-based Epi proColon® test will be examined. Screening eligible average-risk patients identified as non-adherent by medical record will be eligible for the study. Potential subjects will be recruited to participate in a study via mailing and/or at a clinic visit. All study subjects will be enrolled at a clinic visit and will be randomized in two study arms. Those assigned to Arm 1 will be offered a FIT test kit for home use. Those assigned to Arm 2 will be offered a blood draw for the Epi proColon test. Rates of adherence will be compared between those that accept and complete the blood test and those that accept and complete the FIT test. A passive control, usual care arm will comprise subjects meeting eligibility criteria, but not recruited for or participating in the study.

In conjunction with published data (Johnson et al, 2014), the relative utilization of the blood test will be compared to the screening participation via FIT. Increased participation with the Epi proColon blood test could increase screening rates in the non-adherent population. Additionally, for those testing positive in the trial, the rate of adherence to colonoscopy will be determined.

ELIGIBILITY:
Inclusion Criteria:

* 50 years of age or greater, but less than 76 years old
* Has not completed recommended screening for colonoscopy or FIT

  * No colonoscopy in previous 10 years
  * No fecal occult blood test (FOBT) or FIT in previous year and/or > 13 months late FIT
* No flexible sigmoidoscopy in previous 5 years
* Verifiable offer of screening recommendation according to health system standard in at least two independent interactions and a verifiable lack of adherence for two most recent
* Verifiable lack of adherence for >3 months following last screening recommendation
* Primary Care Provider (PCP) has agreed to refer patients for consideration of enrollment in the study
* Subject able to understand and sign written informed consent (IC)

Exclusion Criteria:

* Family history of CRC in a first-degree relative
* Personal history of colonic adenomatous polyps, CRC or inflammatory bowel disease
* Symptoms for which colonoscopy or sigmoidoscopy would otherwise be performed (hematochezia, new onset diarrhea or constipation, abdominal pain)
* Comorbid illness precluding endoscopic evaluation (coronary artery disease with myocardial infarction within 6 months, unstable angina or congestive heart failure, chronic obstructive pulmonary disease requiring home oxygen, other diseases that limit life expectancy to less than 10 years)
* Chronic gastritis, pregnancy, cancer(s) other than colorectal

Ages: 50 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will encompass users of outpatient primary care clinics of one or more health care systems who are considered to be at average-risk for developing colorectal cancer (CRC), have not completed standard screening options, and are not up-to-date with a screening program. Such health care systems may include large healthcare networks with relatively stable patient bases such as Geisinger Health Systems (Danville, PA), Kaiser Permanente (Portland, OR).
Sampling Method: Probability Sample
Enrollment: 490 (Actual)
Dates: Start 2014-10; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Comparison of Adherence to Screening for Each Group | 9 months
  * FIT Test Adherence: Adherence to the FIT Test is expressed as a percentage which is calculated as the number of subjects who complete stool testing within 42 days (6 weeks) divided by the total number of subjects enrolled in the FIT study arm.
  * Epi proColon Test Adherence: Adherence to Epi proColon is expressed as a percentage which is calculated as the number of subjects with documented blood draw for the Epi proColon Test within 42 days (6 weeks) divided by the total number of subjects enrolled in the Epi proColon Test arm.
  * Usual Care Test Adherence: Expressed as a percentage which is calculated as the number of subjects in the Usual Care Group with documented CRC screening (FIT or Colonoscopy) during the duration of the study, divided by the total number of subjects in the usual care group

SECONDARY OUTCOMES:
Adherence to follow-up colonoscopy for tests with a positive result: | 9 months
  Documentation of colonoscopy completed within 42 days (6 weeks) after notification of positive test result
Diagnostic yield of colonoscopy: | 9 months
  Documentation of colonoscopy findings.

CONTACTS AND LOCATIONS:
Overall Officials: Theo deVos, Ph.D., Study Director — Director Development & Commercial Operations
Locations (2):
- United States (2):
  - Kaiser Permanente Center for Health Research, Portland, Oregon
  - Geisinger Clinic, Danville, Pennsylvania

REFERENCES:
- See also: Epigenomics Homepage — http://epigenomics.com